CLINICAL TRIAL: NCT04602143
Title: Therapeutic Effect of Prolonged Testosterone Pretreatment in Women With Poor Ovarian Response: a Randomized Control Trial
Brief Title: Effect of Testosterone Pretreatment in POR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hanoi Medical University (Other)
Collaborators: National Hospital of Obstetrics and Gynecology (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: hoangquochuy, MD
Record Dates: First submitted 2020-10-20; First posted 2020-10-26 (Actual); Last update posted 2020-10-26 (Actual); Status verified 2020-10

CONDITIONS: Infertility
MeSH Terms: conditions — Infertility | interventions — Testosterone

STUDY DESIGN:
Who Masked: Participant
Masking Description: participantes are not aware of treatment groups
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (3):
- Testosterone gel 4 weeks (Experimental): Patients with low ovarian reserve received 4-week TTG application before controlled ovarian hyperstimulation.
  Interventions: Drug: Testosterone gel
- Testosterone gel 6 weeks (Experimental): Patients with low ovarian reserve received 6-week TTG application before controlled ovarian hyperstimulation.
  Interventions: Drug: Testosterone gel
- Control group (No Intervention): Patients with low ovarian reserve received no medication before controlled ovarian hyperstimulation.

INTERVENTIONS:
Drug: Testosterone gel — Apply 12.5mg testosterone gel to the abdomen and rub on with one finger, once a day, in the morning, then allow sites to dry and cover with clothing. Continue the treatment for 4 or 6 weeks until next IVF treatment.
  Other Names: Androgel 1% Transdermal Gel
  Arms: Testosterone gel 4 weeks; Testosterone gel 6 weeks

SUMMARY:
This study compared the therapeutic effect of 4- and 6-week TTG application before controlled ovarian hyperstimulation (COH) in POR.

DETAILED DESCRIPTION:
This randomized control trial (RCT) was conducted between January 2018 and September 2019 at the National Center for Reproductive Medicine, Hanoi, Vietnam. The eligibility of a total of 165 women with POR, undergoing IVF treatment, to be enrolled in the study was assessed. Inclusion criteria included patients who met at least two of the following criteria: (i) having one previous IVF/ intracytoplasmic sperm injection (ICSI) cycle with ≤ 3 oocytes recruited; (ii) AFC ≤ 5-7; and (iii) anti-Mullerian hormone (AMH) ≤ 0.5 - 1.1 ng/mL were enrolled. Exclusion criteria included donated gamete IVF cycles, thyroid disease, liver and kidney dysfunction, and abnormal genitalia. After screening, eligible patients were randomly allocated into two TTG intervention groups (4-week and 6-week groups) and one control group through a manual lottery. Allocation concealment was by sequentially numbered, opaque, sealed envelopes. All participants were blinded to group assignment, but researchers were not blinded.

Serum testosterone are measured before treatment. Durations of androgen supplement are 4 or 6-weeks. After completing the pretreatment, patients are asked to come back when they have menses to begin IVF treatment. Serum testosterone is measured again after the pretreatment in both groups. Patients will be interviewed for side effects and compliance of treatment.

After treatment, patients in both group undergo IVF treatment. IVF treatment will then be performed for all patients, according to the current hospital treatment protocols.

Patients will be followed up at least until 12th week of gestation, if they have positive pregnancy test after embryo transfer.

Data were analyzed using STATA software version 14.0 (Stata Corporation, College Station, TX, USA). Data were analyzed on an intention-to-treat basis. Proportions, means, and standard deviations (SDs) were examined and presented for selected baseline variables by treatment group. Comparisons of baseline characteristics and outcomes by treatment group were performed with the use of ANOVA for continuous variables and a chi-square test for proportions. A Bonferroni correction was used for multiple testing, in which the resulting P-value was multiplied by the number of tests that measured similar constructs. Multivariable logistic regressions were used to quantify the effects of the treatment group, adjusted for all potential confounders including maternal age, body mass index (BMI), infertility duration, primary or secondary infertility, and history of IVF treatment. All statistical tests were two-sided, and P values < 0.05 were considered statistically significant.

ELIGIBILITY:
Inclusion Criteria: patients who met at least two of the following criteria

* Having one previous IVF/ intracytoplasmic sperm injection (ICSI) cycle with ≤ 3 oocytes recruited.
* AFC ≤ 5 - 7.
* Anti-Mullerian hormone (AMH) ≤ 0.5 - 1.1 ng/mL.

Exclusion Criteria:

* donated gamete IVF cycles
* Thyroid disease
* Liver and kidney dysfunction
* Abnormal genitalia

Ages: 20 Years to 47 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 165 (Actual)
Dates: Start 2018-02-16 (Actual); Primary Completion 2020-06-30 (Actual); Study Completion 2020-06-30 (Actual)

PRIMARY OUTCOMES:
Number of oocytes retrieved | 30 minutes after oocyte retrieval complete
  The main outcomes of our study were the total number of retrieved

SECONDARY OUTCOMES:
Pregnancy rates. | 14 days after embryo transfer
  Pregnancy was defined as positive when the serum beta-hCG level was ≥ 50 IU/L
clinical pregnancy rates. | 4 weeks after embryo transfer
  Clinical pregnancy was defined as the presence of a gestational sac identified by transvaginal ultrasound
Ongoing pregnancy rates | after 12 weeks of gestation
  Ongoing pregnancy was defined as a viable intrauterine pregnancy after 12 weeks of gestation.

CONTACTS AND LOCATIONS:
Overall Officials: Hung S Ho, MD, PhD, Study Director — Hanoi Medical University; Tien V Nguyen, MD, PhD, Study Chair — Hanoi Medical University
Locations (1):
- Hanoi Medical University, Vietnam, Hanoi, Vietnam

IPD SHARING:
Plan to Share IPD: No